CLINICAL TRIAL: NCT05159648
Title: Pre-operative, Multi-sensory ICU Simulation Experience to Reduce Post-operative Delirium in the Cardiothoracic Surgical Population
Brief Title: A Study to Evaluate ICU Simulation Experience in the Cardiothoracic Surgical Population to Reduce Post-operative Delirium
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert (Bobby) J. Anderson, Principal Investigator, Mayo Clinic
Other Study IDs: 19-008071
Record Dates: First submitted 2021-10-13; First posted 2021-12-16 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Post-Operative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the effect of a pre-ICU admission virtual reality ICU simulation on post-operative delirium in the elective cardiothoracic surgical population while in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Baseline normal neurological function pre-operatively.
* Planned use of mechanical ventilator with endotracheal tube post-operatively after planned cardiothoracic surgical procedure.

Exclusion Criteria:

* Chronic dementia, Alzheimer's disease, or other chronic neurological disease (i.e., Bi-Polar).
* Chronic use of neurological altering medications such as benzodiazepines, psychotropic, anti-depressants, anxiolytics.
* Patient undergoing emergent surgery.
* Use of post-operative cardiopulmonary support devices such as ECMO (extracorporeal membrane oxygenation), intra-aortic balloon pump, total artificial heart, or other similar device.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with normal neurologic function scheduled for elective cardiothoracic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Anderson, APRN, CNP, DNP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Historical Control Group: Use of standard ultrasound probe for arterial line placement.
- Intervention Group: Use of dual-view ultrasound probe for arterial line placement.
Period: Overall Study
Arm/Group | Historical Control Group | Intervention Group
Started | 139 | 95
Completed | 94 | 44
Not Completed | 45 | 51

BASELINE CHARACTERISTICS:
Groups:
- Historical Control Group: Use of standard single-view ultrasound probe for arterial line placement.
- Total: Total of all reporting groups
Arm/Group | Historical Control Group | Intervention Group | Total
Number analyzed (Participants) | 139 | 95 | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 139 | 95 | 234
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 72 [65 to 77] | 50 [42 to 58] | 60 [42 to 77]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender information was only collected from subjects who completed the study
  Participants
    number analyzed (Participants) | 94 | 44 | 138
    Female | 22 | 10 | 32
    Male | 72 | 34 | 106
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 139 | 95 | 234
Neurocognitive disorder [Count of Participants; unit: Participants] | 106 | 95 | 201
Use of neurologic altering medication [Count of Participants; unit: Participants] | 131 | 95 | 226
Return to operating room prior to discharge from ICU [Count of Participants; unit: Participants] | 135 | 95 | 230

OUTCOME MEASURES:

1. Primary Outcome: Confusion Assessment Method for the ICU (CAM-ICU)
Description: Number of Participants with one or more Positive Confusion Assessment. "Confusion Assessment Method for the ICU" - Establishes ability to detect delirium in high-risk settings such as the intensive care unit. Recorded during every scheduled patient assessment by nurse and with mental changes. Reports as "Positive" or "Negative" with response to different assessments regarding level of consciousness, acute onset or fluctuating course of mental status and inattention.
Time Frame: Once, during ICU admission within 24 hours of ICU admission.
Measure: Count of Participants; unit: Participants
Groups:
- Historical Control Group: Routine post operative intensive care unit care.
- Intervention Group: Pre-operative virtual reality simulation.
Arm/Group | Historical Control Group | Intervention Group
Number analyzed (Participants) | 94 | 44
Participants | 4 | 1

2. Primary Outcome: Subjective Experiential Outcome After ICU Simulation
Description: Survey questions to understand patient's subjective experience during the virtual reality ICU simulation session. Internally created survey. The number of subjects who completed the survey.
Time Frame: Once, immediately following the virtual reality ICU simulation session.
Population: Data was not collected nor analyzed for 68 subjects in the control group as they chose not to complete the survey.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: Patients exposed to pre-operative virtual reality simulation.
Arm/Group | Historical Control Group | Intervention Group
Number analyzed (Participants) | 94 | 44
Participants | 26 | 44

3. Primary Outcome: Subjective Experiential Outcome After ICU Admission
Description: Survey questions to understand patient's subjective experience in the intensive care unit. The number of subjects who completed the survey.
Time Frame: Once, up to 3 days after transfer out of the Intensive Care Unit.
Population: Data was not collected nor analyzed for 68 subjects in the control group as they chose not to complete the survey.
Measure: Count of Participants; unit: Participants
Groups:
- Historical Control Group: Standard post-operative care in the intensive care unit.
Arm/Group | Historical Control Group | Intervention Group
Number analyzed (Participants) | 94 | 44
Participants | 26 | 44

4. Secondary Outcome: Duration of ICU Admission
Description: Number of hours in the intensive care unit measured in the electronic health record from admission time to the ICU to discharge time from the ICU.
Time Frame: During ICU admission; average 2 days
Reporting Status: Not Posted

5. Secondary Outcome: Duration of Intravenous Sedation in the ICU
Description: Number of hours of intravenous sedation in the ICU measured through the medication administration record via the electronic healthcare record.
Time Frame: During ICU admission; average 2 days
Reporting Status: Not Posted

6. Secondary Outcome: Duration of Mechanical Ventilation in the ICU
Description: Number of hours of mechanical ventilation in the ICU measured via the electronic healthcare record with data imported into the electronic healthcare record directly from the mechanical ventilator.
Time Frame: During ICU admission; average 2 days
Reporting Status: Not Posted

7. Secondary Outcome: Use of Anti-psychotic Medications
Description: Number of antipsychotic medication administrations in the ICU measured through the medication administration record via the electronic healthcare record.
Time Frame: Throughout ICU admission; average of 5 days
Reporting Status: Not Posted

8. Secondary Outcome: Cardiopulmonary Bypass
Description: Number of hours of use of cardiopulmonary bypass in the operating room via record from the cardiopulmonary bypass perfusionist in the operating room imported into the electronic healthcare record.
Time Frame: During OR case; average 12 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events will be collected for all participants from baseline to end of study, approximately five days
Arm/Group | Historical Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/95
Other Adverse Events (participants affected / at risk) | 0/139 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT05159648/Prot_000.pdf